CLINICAL TRIAL: NCT01049997
Title: Frailty as an INstrument for Evaluation of Elderly Patients With Non ST Elevation Myocardial Infarction (NSTEMI)
Acronym: FINE75+
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Niklas Ekerstad, MD,PhD, Linkoeping University
Other Study IDs: FINE75+
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Non ST Elevation Myocardial Infarction (NSTEMI); Frailty
Keywords: Non ST Elevation Myocardial Infarction (NSTEMI); Elderly; Frailty
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NSTEMI75+: Patients, 75 years old or older, with Non ST Elevation Myocardial Infarction (NSTEMI)

SUMMARY:
The purpose of this study is to describe patients, 75 years old or older, with Non ST Elevation Myocardial Infarction (NSTEMI) especially regarding the following variables: cardiovascular risk, co-morbidity and frailty. The investigators hypothesize that the degree of frailty influences the benefit from coronary angiography and the possible invasive treatment which can follow.

DETAILED DESCRIPTION:
The term frailty denotes a multi-dimensional syndrome characterized by increased vulnerability and decreased physiologic reserves. Frailty stratification predicts a patient's risk of death and need for institutional care. The construct is well validated, but there is not one single accepted operational definition. The CSHA Clinical Frailty Scale (CFS) is a 7-point scale relying on clinical judgement. It is a global clinical measure of biological age, and it mixes co-morbidity, disability and cognitive impairment.Though frailty instruments so far mainly have been used in a geriatric context, it has been pointed out as relevant for cardiologic patients as well, e.g. regarding risk stratification for elderly patients with NSTEMI. The purpose of this study is to describe patients, 75 years old or older, with Non ST Elevation Myocardial Infarction (NSTEMI) especially regarding the following variables: cardiovascular risk, co-morbidity and frailty. The investigators hypothesize that the degree of frailty influences the benefit from coronary angiography and the possible invasive treatment which can follow.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 75 years old or older, with diagnosed NSTEMI, and cared for at one of the following hospital care units: cardiology, acute medicine, geriatrics, other internal medicine unit.

Exclusion Criteria:

* Not willing to participate.
* Non-evaluable patient due to communication problems and insufficient clinical information for the judgement of frailty (CFS).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive evaluable patients, 75 years old or older, with diagnosed NSTEMI, and cared for at one of the following hospital care units in the University Hospital of Linköping and the County Hospitals in Trollhättan (NÄL-Uddevalla) and Jönköping (Ryhov): cardiology, acute medicine, geriatrics, other internal medicine unit.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The composite of death from any cause, myocardial infarction, revascularization due to ischemia, hospitalization from any cause, major bleeding, stroke/TIA and need for dialysis by one month after inclusion. | One month after inclusion

SECONDARY OUTCOMES:
The composite of major bleeding, stroke/TIA and need for dialysis by one month after inclusion. | One month after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Niklas G Ekerstad, MD, Principal Investigator — Linkoeping University, Sandbäcksgatan 7, 58183 Linkoeping, Sweden; Joakim Alfredsson, PhD, Principal Investigator — Department of Cardiology, University Hospital of Linkoeping, 58183 Linkoeping, Sweden; Marcus Lindenberger, PhD, Principal Investigator — Department of Cardiology, County Hospital Ryhov, 551 85 Joenkoeping, Sweden
Locations (1):
- The Center for Medical Technology Assessment/IMH, Linkoeping University, Linköping, Östergötland County, Sweden